CLINICAL TRIAL: NCT02701244
Title: A Multicenter Registry Study of Breast Microseed Treatment for Early Stage Breast Cancer
Brief Title: A Registry Study of Breast Microseed Treatment
Status: Recruiting | Type: Observational
Sponsor: Concure Oncology-Breast Microseed Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BMS-001
Record Dates: First submitted 2016-02-25; First posted 2016-03-08 (Estimated); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Breast Neoplasms
Keywords: Infiltrating Ductal Carcinoma; Ductal Carcinoma In Situ; Brachytherapy; Breast Neoplasms; Breast Diseases; Neoplasms; Neoplasms by Site
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating; Breast Diseases; Neoplasms; Neoplasms by Site

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Permanent Breast Seed Implant (PBSI): Women with eligible early stage breast cancer who received a permanent breast seed implant status post lumpectomy
  Interventions: Radiation: Permanent Breast Seed Implant (PBSI)

INTERVENTIONS:
Radiation: Permanent Breast Seed Implant (PBSI) — Patients are pre-planned using Computerized Tomography (CT) simulation. Implant is performed after surgery under light sedation and local freezing (alternatively general anesthesia). Stranded seeds are inserted using a brachytherapy template that is immobilized to the planned target volume using a 'localization' needle. Patients are released the same day and Quality Assurance involves post-implant Computerized Tomography (CT).
  Other Names: Breast Microseed Treatment

SUMMARY:
For women diagnosed with early stage breast cancer, lumpectomy followed by radiation is a common treatment option. Radiation treatment is typically delivered to the whole breast, five times per week, for anywhere from 3 to 8 weeks. The radiation helps kill any cancer cells that may have been left over following the surgery but causes skin burns. Many studies have demonstrated that radiation to the whole breast is not necessary, that it can be delivered to a portion of the breast where the cancer is more likely to recur.

A technique called a Permanent Breast Seed Implant (PBSI) involving the implantation of radioactive seeds has been developed to deliver the radiation to a portion of the breast. The procedure is performed on an out-patient basis under local anesthesia and light sedation. Because the radioactive seeds are permanently implanted in the breast, the patient is able to live a normal life while the seeds deliver the prescribed radiation to the breast.

Previous studies on PBSI demonstrate that it is a safe and effective alternative form of radiation for appropriately selected patients after lumpectomy. However, those results have been obtained mainly from a single institution, with only 4 patients treated in another center. Further research is still needed to evaluate its safety in a multi-center setting. The purpose of this study is to ensure the appropriate training of clinicians who will be performing this procedure and to capture long term outcomes and rare complications if any.

DETAILED DESCRIPTION:
For women diagnosed with early stage breast cancer, lumpectomy followed by radiation is a common treatment option. Radiation treatment is typically delivered to the whole breast, five times per week, for anywhere from 3 to 8 weeks. The radiation helps kill any cancer cells that may have been left over following the surgery but causes skin burns. Many studies have demonstrated that radiation to the whole breast is not necessary, that it can be delivered to a portion of the breast where the cancer is more likely to recur.

A technique called a Permanent Breast Seed Implant (PBSI) involving the implantation of radioactive seeds has been developed to deliver the radiation to a portion of the breast. The procedure is performed on an out-patient basis under local anesthesia and light sedation. Because the radioactive seeds are permanently implanted in the breast, the patient is able to live a normal life while the seeds deliver the prescribed radiation to the breast.

Previous studies on Permanent Breast Seed Implant (PBSI) demonstrate that it is a safe and effective alternative form of radiation for appropriately selected patients after lumpectomy. However, those results have been obtained mainly from a single institution, with only 4 patients treated in another center. Further research is still needed to evaluate its safety in a multi-center setting. The purpose of this study is to ensure the appropriate training of clinicians who will be performing this procedure and to capture long term outcomes and rare complications if any.

Due to the wide-spread use of mammography, breast cancer is commonly diagnosed at an early stage. The standard treatment for early-stage disease is breast conserving surgery followed by adjuvant radiation therapy to the whole breast. This approach leads to low recurrence rates with a good cosmesis and provides an effective alternative to mastectomy. However, half of these women will develop significant acute skin toxicity following whole breast irradiation. These reactions occur more frequently in the infra-mammary fold, are associated with pain, and are associated with a reduction in health-related quality of life. Whole breast radiotherapy involves several daily treatments delivered over a period of 3 to 7 weeks which can be disruptive for the patient's life.

To address these drawbacks, the concept of accelerated partial breast irradiation was proposed. It arose out of the realization that the majority of tumor recurrences occur at or near the region of the prior lumpectomy site, suggesting that for well selected patients only the breast tissue surrounding the tumor bed might need radiation treatment. Accelerated partial breast irradiation limits the radiation to a smaller portion of the breast (surrounding the tumor cavity) and has the advantages of reducing radiation-induced toxicity at increased convenience because it is delivered within a much shorter period of time. In reducing the volume of breast treated, a higher dose of radiation can be delivered in each treatment session. Accelerated partial breast irradiation advantages include a reduction of the amount of irradiated skin and therefore the possibility to reduce radiation-induced skin toxicity, and an increased convenience because it can be accelerated.

Several accelerated partial breast irradiation techniques have been reported including external beam conformal irradiation, intra-operative radiotherapy and brachytherapy techniques. Brachytherapy has been the most widely evaluated accelerated partial breast irradiation technique. It involves the insertion of radioactive material directly into the surgical cavity using tubes or catheters. Treatments are generally delivered as an outpatient procedure using high dose rate (HDR) brachytherapy, delivering multiple treatments (8 to 10) over a period of 5 to 8 days. Intra-operative radiotherapy is delivered in a single session at the time of initial surgery.

A permanent breast seed implant (PBSI) technique of partial breast irradiation using palladium (103Pd) seeds has been proposed. Similar to a permanent seed implant used to treat prostate cancer, permanent breast seed implant (PBSI) involves the insertion of stranded radioactive seeds under ultra-sound guidance. The advantages of the permanent breast seed implant (PBSI) technique over other brachytherapy techniques include: i/- it is an out-patient procedure performed in a single one-hour session under local anesthesia and light sedation; ii/- it is performed after the surgery when the final pathology report is available and the scar is completely healed; and iii/- the use of a low dose rate technique presents the possible advantage to be more efficient and better tolerated compared to high dose rate techniques.

The local recurrence rate, immediate and delayed toxicity, the radiation safety and quality assurance data suggest that permanent breast seed implant (PBSI) is a safe and acceptable option of accelerated partial breast irradiation, capable of delivering the right amount of dose in the right location for selected early stage breast cancer. However, those results have been obtained mainly from a single institution, with 4 patients treated in another center. Further research is still needed to evaluate its safety in a multi-center setting and also to detect serious adverse events when a larger number of patients are treated by a larger group of practitioners. Since brachytherapy is operator dependent, a registry represents a unique opportunity to ensure the appropriate training of radiation oncologist and to capture capturing long terms outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of invasive or in-situ ductal carcinoma (DCIS)
* Treated by breast conserving surgery with axillary node dissection (with a minimum of 6 nodes sampled) or sentinel lymph node biopsy
* Surgical margins clear for invasive carcinoma (no tumor at ink margin) or superior or equal to 2 mm for in-situ ductal carcinoma (DCIS)
* A maximum tumor size of 3 cm
* Age ≥50 years old
* Informed consent signed if participating in the Registry

Exclusion Criteria:

* No previous cancer unless in remission for more than 2 years.
* Active auto immune disorder with severe vasculitis component
* Uncontrolled and complicated insulin-dependent diabetes
* Pregnancy
* Cosmetic breast implants
* Psychiatric or addictive disorder that would preclude attending follow-up
* Post-operative breast infection requiring prolonged antibiotic therapy
* Lobular features on histology (pure or mixed) or sarcoma histology
* Node macroscopically positive on axillary dissection or in the sentinel lymph node biopsy
* Extensive in- situ carcinoma
* Multicentric disease (in more than one quadrant or separated by 2 cm or more)
* Paget's disease of the nipple
* Metastases
* Patients presenting with a large post-surgical fluid cavity as determined on the planning Ultrasound (US), resistant to the application of hot compresses for 4 weeks
* Clear delineation of the target volume on Computerized Tomography (CT) is not possible
* Volume to be implanted over 150cc
* Target volume too close to skin such that the 90% isodose overlaps the skin surface

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are identified during a new patient consult in each participating center.
Sampling Method: Non-Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2016-07; Primary Completion 2021-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Serious Adverse Events (SAE) | Up to 10 years from procedure date
  Serious Adverse Events (SAE) is an unintended sign, symptom, or syndrome illness that occurs during the period of observation in the clinical study and that is life threatening or result in death. Serious Adverse Events (SAE) corresponds to grade 4 or 5 signs or symptoms from the National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) version 4.03 scale.

SECONDARY OUTCOMES:
Breast Cancer Recurrence | Up to 10 years from procedure date
  Ipsilateral in-breast or chest wall recurrence is defined as evidence of invasive or in situ breast cancer (except lobular carcinoma in-situ (LCIS)) in the ipsilateral breast. It is important to get a pathology confirmation of the recurrence.
  In case of ipsilateral recurrence or second primary breast cancer, a copy of the clinic note summarizing the localization (same quadrant, other quadrant, not specified), the pathology, the work-up and treatment plan will be submitted to the Registry. Patients will be followed beyond the diagnosis for survival assessment.
Permanent Breast Seed Implant (PBSI) Side Effects | At 2 months from procedure date
  Any toxicity related to the radiation treatment, including skin and subcutaneous, or any other organ in case of seed migration will be coded using the National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) version 4.03 scale.
Permanent Breast Seed Implant (PBSI) Side Effects | Yearly up to 10 years from procedure date
  Any toxicity related to the radiation treatment, including skin and subcutaneous, or any other organ in case of seed migration will be coded using the National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) version 4.03 scale.
Cosmetic Outcome | Yearly up to 10 years from procedure date
  Cosmetic results will be self-evaluated at each follow-up visit by the patients using the Breast Cancer Treatment Outcome Scale (BCTOS) questionnaire
Survival (either free of cancer or with disease present) | Up to 10 years from procedure date
  Patient survival, either free of cancer or with disease present will be recorded at follow-up appointments

CONTACTS AND LOCATIONS:
Overall Officials: Juanita Crook, MD, Principal Investigator — British Columbia Cancer Agency; Jean-Philippe Pignol, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (3):
- United States (3):
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Mary Washington Hospital, Fredericksburg, Virginia
  - Swedish Cancer Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pignol JP, Rakovitch E, Keller BM, Sankreacha R, Chartier C. Tolerance and acceptance results of a palladium-103 permanent breast seed implant Phase I/II study. Int J Radiat Oncol Biol Phys. 2009 Apr 1;73(5):1482-8. doi: 10.1016/j.ijrobp.2008.06.1945. Epub 2008 Oct 18. PMID 18930602
- [Background] Pignol JP, Caudrelier JM, Crook J, McCann C, Truong P, Verkooijen HA. Report on the Clinical Outcomes of Permanent Breast Seed Implant for Early-Stage Breast Cancers. Int J Radiat Oncol Biol Phys. 2015 Nov 1;93(3):614-21. doi: 10.1016/j.ijrobp.2015.07.2266. Epub 2015 Jul 21. PMID 26461003
- [Background] Pignol JP, Keller B, Rakovitch E, Sankreacha R, Easton H, Que W. First report of a permanent breast 103Pd seed implant as adjuvant radiation treatment for early-stage breast cancer. Int J Radiat Oncol Biol Phys. 2006 Jan 1;64(1):176-81. doi: 10.1016/j.ijrobp.2005.06.031. Epub 2005 Sep 22. PMID 16182464
- [Background] Keller BM, Pignol JP, Rakovitch E, Sankreacha R, O'Brien P. A radiation badge survey for family members living with patients treated with a (103)Pd permanent breast seed implant. Int J Radiat Oncol Biol Phys. 2008 Jan 1;70(1):267-71. doi: 10.1016/j.ijrobp.2007.08.006. Epub 2007 Oct 29. PMID 17967512
- [Background] Keller B, Sankreacha R, Rakovitch E, O'brien P, Pignol JP. A permanent breast seed implant as partial breast radiation therapy for early-stage patients: a comparison of palladium-103 and iodine-125 isotopes based on radiation safety considerations. Int J Radiat Oncol Biol Phys. 2005 Jun 1;62(2):358-65. doi: 10.1016/j.ijrobp.2004.10.014. PMID 15890575